CLINICAL TRIAL: NCT00791440
Title: Psychosis in Schizophrenia: Mechanisms of Recovery
Brief Title: Recovery From Psychosis in Schizophrenia - The Impact of Cognitive-Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5808; K23MH077653 (NIH)
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Schizoaffective; Schizophreniform; Psychosis; Psychotic; Hallucinations; Delusions; Paranoia; Paranoid; Voices; CBT; Cognitive Behavior Therapy; Cognitive Therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders; Hallucinations; Delusions; Paranoid Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Up to 26 sessions (over a 30 week period) of weekly, individual Cognitive-Behavior Therapy (CBT) to target hallucinations and delusions in addition to standard psychiatric treatment.
  Interventions: Behavioral: Cognitive-Behavior Therapy
- 2 (Active Comparator): 30 weeks of standard psychiatric treatment.
  Interventions: Other: Standard Psychiatric Treatment

INTERVENTIONS:
Behavioral: Cognitive-Behavior Therapy — Weekly individual Cognitive-Behavior Therapy (CBT) to target hallucinations and delusions in addition to standard psychiatric treatment.
  Other Names: CBT for psychosis
  Arms: 1
Other: Standard Psychiatric Treatment — Standard psychiatric treatment.
  Other Names: Treatment As Usual (TAU)
  Arms: 2

SUMMARY:
This study examines the impact of Cognitive-Behavior Therapy (CBT) on symptoms, physiological arousal, stressors, and the ways to deal with them in individuals with schizophrenia and related disorders. The primary aim of this study is to investigate the role cognitive coping strategies play in mediating the link between stress, physiological arousal, and psychotic symptoms in individuals with schizophrenia during recovery from psychosis.

DETAILED DESCRIPTION:
This study examines the mechanisms of recovery from psychosis. Specifically, the study aims to evaluate the putative impact of enhancing cognitive coping strategies via Cognitive-Behavior Therapy for psychosis (CBTp) on subjective stress, autonomic regulation (physiological arousal), and psychotic symptoms in individuals with schizophrenia and related disorders. As part of the study, participants will be randomized to receive up to 26 weekly sessions of CBTp (over 30 weeks) or "treatment as usual". Research evaluations will completed at baseline, and after 10, 20 and 30 weeks. The study outcome measures include psychotic symptoms as measured by clinical interviews, along with ambulatory measures of autonomic regulation and self-reports of psychotic experiences during daily functioning using mobile devices (i.e., Palm computers).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages 18-50.
* Have capacity to give informed consent.
* English speaking.
* Have a DSM-IV diagnosis of schizophrenia, or schizoaffective disorder, or schizophreniform disorder.
* Presence of active psychosis as indexed by ratings ≥3 on any hallucinations and delusions items of the Scale for Assessment of Positive Symptoms (SAPS).

Exclusion Criteria:

* Lacks capacity to give informed consent.
* Diagnosis of mental retardation (IQ < 80).
* Have history of neurological disorders or medical conditions known to seriously affect the brain.
* Have history of cardiac conditions or hypertension; current use of anti-cholinergic, beta-blockers, anti-histamine, or anti-hypertensive medication; abnormalities on ECG.
* Have used street drugs within the past 4 weeks.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment of Positive Symptoms (SAPS) | At Baseline and after 10, 20 and 30 weeks

SECONDARY OUTCOMES:
Momentary self-report ratings of psychotic symptoms using a Palm computer | At Baseline and after 30 weeks
Momentary self-report ratings of stress and coping strategies using a Palm computer | at Baseline and after 30 weeks
Momentary ambulatory measures of heart rate and breathing | At Baseline and after 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Kimhy, Ph.D., Principal Investigator — Columbia University & New York State Psyciatric Institute
Locations (1):
- Columbia University & New York State Psyciatric Institute, New York, New York, United States